CLINICAL TRIAL: NCT05029141
Title: A Multi-center, Randomized Clinical Trial of Chidamide Combined With Azacytidine and the HAG Regimen in the Treatment of Relapsed/Refractory Acute Myeloid Leukemia Patients
Brief Title: New Double Epigenetic Regimen in the Treatment of Relapsed or Refractory Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Ruijin Hospital (Other); West China Hospital (Other); Fujian Medical University Union Hospital (Other); The First Hospital of Jilin University (Other); Anhui Provincial Hospital (Other Government); Qilu Hospital of Shandong University (Other); The Affiliated Cancer Hospital of Zhengzhou University (Unknown); Shandong Provincial Hospital (Other Government); Nanfang Hospital, Southern Medical University (Other); First Affiliated Hospital of Harbin Medical University (Other); Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Sheng-Li Xue, MD, accociate professor, The First Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZCAHAG
Record Dates: First submitted 2021-08-16; First posted 2021-08-31 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukemia; Refractory Acute Leukemia; Relapsed Adult AML
Keywords: chidamide; Azacitidine; priming regimen
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chidamide+AZA+HHT+AraC+G-CSF group (Experimental): The patients are randomized into the group. Patients whose last induction failure regimen is a demethylated agent combined with priming regimen enter the experimental group directly.
  Interventions: Drug: CAHAG regimen
- Placebo+AZA+HHT+AraC+G-CSF group (Placebo Comparator): The patients are randomized into the group.
  Interventions: Drug: Placebo regimen

INTERVENTIONS:
Drug: CAHAG regimen — Chidamide 30mg orally twice every week for 2 weeks on days 1, 4, 8, 11, azacytidine 75mg/m2 intravenously daily for 7 days (d3-d9) and HAG regimen (cytarabine, 10 mg/m2 subcutaneously every 12 h on days 3-16; homoharringtonine, 1mg/m2 intravenously every day on days 3-16; and concurrent granulocyte colony-stimulating factor, 200mg/m2/day subcutaneously daily from days 2 to neutral granulocyte recovery. (when WBC > 20×10E9/L, G-CSF paused).
  One treatment cycle for 28 days, a total of 2 cycles. If the bone marrow assessment is MLFS on the 28th day in the first cycle, the second cycle of treatment will be started after NE<1.0×10E9/L; if the delay exceeds 2 weeks, the patient needs to withdraw from the trial.
  Arms: Chidamide+AZA+HHT+AraC+G-CSF group
Drug: Placebo regimen — Chidamide 0mg orally twice every week for 2 weeks on days 1, 4, 8, 11, azacytidine 75mg/m2 intravenously daily for 7 days (d3-d9) and HAG regimen (cytarabine, 10 mg/m2 subcutaneously every 12 h on days 3-16; homoharringtonine, 1mg/m2 intravenously every day on days 3-16; and concurrent granulocyte colony-stimulating factor, 200mg/m2/day subcutaneously daily from days 2 to neutral granulocyte recovery. (when WBC > 20×10E9/L, G-CSF paused).
  One treatment cycle for 28 days, a total of 2 cycles. If the bone marrow assessment is MLFS on the 28th day in the first cycle, the second cycle of treatment will be started after NE<1.0×10E9/L; if the delay exceeds 2 weeks, the patient needs to withdraw from the trial.
  Arms: Placebo+AZA+HHT+AraC+G-CSF group

SUMMARY:
This study is to investigate the therapeutic efficacy and side effect of chidamide, azacitidine combined with priming HAG regimen for relapsed or refractroy acute myeloid leukemia

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 and ≤ 70 years
* Patients diagnosed with AML according to 2016 WHO myeloid malignant disease diagnosis standard (Non-APL)
* Patients with AML must meet one of the following criteria, A or B:

A: Refractory AML disease was defined as follows: (1) failure to attain CR following exposure to at least 2 courses of standard or intensive induction therapy; or (2) bone marrow leukemia cell decline index (BMCDI) < 50% and > 20% after 1 course of standard or intensive induction therapy. B: Relapsed AML disease was defined as follows: (1) reappearance of leukemic blasts in the peripheral blood after CR; or (2) detection of ≥ 5% blasts in the BM not attributable to another cause (e.g., BM regeneration after consolidation therapy); or (3) extramedullary relapse.

* ECOG performance status score less than 3
* Expected survival time ˃ 3 months
* Patients without serious heart, lung, liver, or kidney disease
* Ability to understand and voluntarily provide informed consent

Exclusion Criteria:

* Patients who are allergic to the study drug or drugs with similar chemical structures
* Pregnant or lactating women, and women of childbearing age who do not want to practice effective methods of contraception
* Active infection
* Active bleeding
* Patients with new thrombosis, embolism, cerebral hemorrhage, or other diseases or a medical history within one year before enrollment
* Patients with mental disorders or other conditions whereby informed consent cannot be obtained and where the requirements of the study treatment and procedures cannot be met
* Liver function abnormalities (total bilirubin > 1.5 times the upper limit of the normal range, ALT/AST > 2.5 times the upper limit of the normal range or patients with liver involvement whose ALT/AST > 1.5 times the upper limit of the normal range), or renal anomalies (serum creatinine > 1.5 times the upper limit of the normal value)
* Patients with a history of clinically significant QTc interval prolongation (male > 450 ms; female > 470 ms), ventricular heart tachycardia and atrial fibrillation, II-degree heart block, myocardial infarction attack within one year before enrollment, and congestive heart failure, and patients with coronary heart disease who have clinical symptoms and requiring drug treatment
* Surgery on the main organs within the past six weeks
* Drug abuse or long-term alcohol abuse that would affect the evaluation results
* Patients who have received organ transplants (excepting bone marrow transplantation)
* Patients not suitable for the study according to the investigator's assessment

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | At the end of Cycle 1 (each cycle is 28 days)
  The overall response (completed remission without minimal residual disease, completed remission with incomplete blood count recovery, morphologic leukemia-free state and partial remission) rate achieved after one or two courses(28 days) induction therapy by CAHAG regimen.
Complete remission without minimal residual disease (CR with MRD-) | At the end of Cycle 1 (each cycle is 28 days)
  If studied pretreatment, CR with negativity for a genetic marker by RT-qPCR, or CR with negativity by MFC
Complete remission with incomplete hematologic recovery (CRi) | At the end of Cycle 1 (each cycle is 28 days)
  All CR criteria except for residual neutropenia (,1.0*10E9/L [1000/uL]) or thrombocytopenia (<100*10E9/L [100 000/uL])
Morphologic leukemia-free state (MLFS) | At the end of Cycle 1 (each cycle is 28 days)
  Bone marrow blasts ,5%; absence of blasts with Auer rods; absence of extramedullary disease; no hematologic recovery required
Partial remission (PR) | At the end of Cycle 1 (each cycle is 28 days)
  All hematologic criteria of CR; decrease of bone marrow blast percentage to 5% to 25%; and decrease of pretreatment bone marrow blast percentage by at least 50%.

SECONDARY OUTCOMES:
Duration of Response (DOR) | 1 year
  It is measured the time from initial response to subsequent disease progression or relapse.
Overall Survival (OS) | 1 year
  It is measured from the time of entry into this trial to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.
Progression-Free Survival (PFS) | 1 year
  It is measured from the time from randomization to progression or death.

OTHER OUTCOMES:
Adverse reactions in hematology | At the end of Cycle 1 (each cycle is 28 days)
  Record of adverse events in hematological system during and after CAHAG regimen induction (agranulocytosis days, PLT/RBC transfusion units).
Nonhematological adverse reactions | At the end of Cycle 1 (each cycle is 28 days)
  Record of adverse events in other organs or systmes during and after CAHAG regimen induction (infection and organ injury).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No